CLINICAL TRIAL: NCT05409833
Title: Systemic Transthyretin Amyloidosis: Carpal Tunnel Syndrome in a Portuguese Population (CarPoS Study)
Brief Title: Systemic Transthyretin Amyloidosis: Carpal Tunnel Syndrome in a Portuguese Population
Acronym: CarPoS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar De São João, E.P.E. (Other); Centro de Investigação em Tecnologias e Serviços de Saúde (Other); Rede de Investigação em Saúde (Other)
Responsible Party: Sponsor
Other Study IDs: CarPoS
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-06

CONDITIONS: Transthyretin Amyloidosis; Carpal Tunnel Syndrome
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — biopsy and peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Patients aged ≥ 60 years old with symptomatic carpal tunnel syndrome submitted to surgery
  Interventions: Diagnostic Test: Synovial biopsy and Cardiac scintigraphy with [99mTc]Tc-DPD
- Group 2: Patients aged ≥ 60 years old without symptomatic carpal tunnel syndrome submitted to hand surgery
  Interventions: Diagnostic Test: Synovial biopsy and Cardiac scintigraphy with [99mTc]Tc-DPD

INTERVENTIONS:
Diagnostic Test: Synovial biopsy and Cardiac scintigraphy with [99mTc]Tc-DPD — Congo red and Immunohistochemical analysis and/or Mass spectrometry analysis

SUMMARY:
Systemic transthyretin amyloidosis is an aging-related disorder. It is usually associated with cardiac disease but also extends to other organs. Recent studies found that idiopathic carpal tunnel syndrome patients may have amyloid deposition in tenosynovial tissue. The main aims of this project are the characterization of the association between idiopathic carpal tunnel syndrome and transthyretin amyloidosis and its evaluation as a predictive factor of cardiac amyloidosis

ELIGIBILITY:
Inclusion Criteria:

. Patients aged ≥ 60 years old with symptomatic idiopathic carpal tunnel syndrome or other hand surgery indications.

Exclusion Criteria:

. Diabetes mellitus, hypothyroidism, hemodialysis, rheumatoid arthritis, and other inflammatory arthropathies, multiple myeloma, gout, chondrocalcinosis, Colles fracture, space-occupying lesions, and infectious synovitis.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ≥60 years old submitted to hand surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of transthyretin amyloidosis in synovial in patients with ≥60 years old | 24 months
  Number of patients with transthyretin amyloidosis in synovial in relation to total number of patients submitted to hand surgery

SECONDARY OUTCOMES:
Association between synovial transthyretin amyloidosis with carpal tunnel syndrome | 24 months
  Comparison between group 1 and 2
Association between idiopathic carpal tunnel syndrome with cardiac transthyretin amyloidosis | 24 months
  Comparison between group 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Elisabete Martins, MD, PhD, Principal Investigator — Universidade do Porto
Locations (2):
- Portugal (2):
  - Centro Hospitalar Universitário São João, Porto
  - Faculty of Medicine (FMUP), Porto